CLINICAL TRIAL: NCT02389023
Title: Multicenter, Prospective, Randomized Clinical Trial of a Negative Pressure Incision Management System in High Risk Vascular Surgery Patients
Brief Title: Comparison of Prevena Negative Pressure Incision Management System vs. Standard Dressing After Vascular Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont Medical Center (Other)
Collaborators: KCI USA, Inc (Industry); MaineHealth (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Bertges, MD, Vascular Surgeon, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15371
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Peripheral Artery Disease; Critical Limb Ischemia; Claudication
Keywords: surgical site infection; infrainguinal bypass; incisional wound vacuum assisted closure; Prevena
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Intermittent Claudication; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard gauze dressing (Other): a standard post-operative dressing consisting of dry gauze and tape will be placed over the surgical site
  Interventions: Other: standard gauze dressing
- Prevena Incision Management System (Other): the Prevena™ Incision Management System (PIMS) or ActiVAC® with the PrevenaTM Dressings (Peel and Place™ or Customizable™) will be placed over the surgical site. The Prevena dressing is not considered experimental and has FDA approval for coverage of at risk closed-surgical incisions. The dressing is already in clinical use for vascular surgery bypass operations at the University of Vermont Medical Center.
  Interventions: Other: Prevena Incision Management system

INTERVENTIONS:
Other: standard gauze dressing — Standard gauze dressing with tape will be placed over the surgical incision in the operating room and left on the incision as dictated by standard of care
  Arms: standard gauze dressing
Other: Prevena Incision Management system — The Prevena dressing system over the closed surgical incision. The dressing consists of a sterile sponge that is placed over the incision followed by a plastic adhesive covering that is used to secure it to the skin forming an air-tight seal. The sponge is then connected by tubing to a vacuum that applies negative pressure to the closed system. This allows fluid to drain from the wound and into a container connected to the dressing.
  Arms: Prevena Incision Management System

SUMMARY:
The purpose of this study is to evaluate the effectiveness of negative pressure incision management system (Prevena™ Incision Management System (PIMS) or ActiVAC® with the Prevena™ Dressings (Peel and Place™ or Customizable™), KCI) in the prevention of wound complications including surgical site infection (SSI) and non-infectious complications in patients undergoing vascular surgery with groin incisions.

DETAILED DESCRIPTION:
Complications such as surgical site infections, deep wound infections, prosthetic graft infections, and non-infections problems such as wound dehiscence continue to cause significant morbidity for patients undergoing arterial reconstruction for peripheral arterial disease. Patients undergoing leg bypass surgery for limb salvage are at particular risk due to their medical problems such as diabetes and renal failure and location of incisions along the groin area. Surgical site infections (SSI) are estimated to occur in 5-40% of patients undergoing arterial bypass for lower extremity arterial occlusive disease. The in-hospital SSI rate is 5% across the Vascular Study Group of New England, a regional quality improvement registry. Factors contributing to wound infections include patient factors such as advanced age and comorbidities such as obesity, diabetes and renal insufficiency and surgical factors including the division of local lymphatics in the groin, placement of a prosthetic graft and inherent difficulty in keeping an incision across the groin crease covered, dry and protected.

Despite the use of standard sterile technique and perioperative preventative antibiotics infections these complications continue to cause patient morbidity. In addition these complications increase the intensity and cost of care with an added estimated expense of $11,000 per incident. New strategies are needed to reduce these complications. Negative pressure wound therapy has the potential to prevent a variety of wound complications. One innovative strategy that has shown promise is the application of the Prevena dressing system over the closed surgical incision. The dressing consists of a sterile sponge that is placed over the incision followed by a plastic adhesive covering that is used to secure it to the skin forming an air-tight seal. The sponge is then connected by tubing to a vacuum that applies negative pressure to the closed system. This allows fluid to drain from the wound and into a container connected to the dressing. When compared to surgical dressing with sterile gauze and tape, the Prevena dressing system has the advantages of providing a sterile barrier, reducing tension on the incision, and removing fluid from the incision. Please refer to patient brochure for an illustration and further description of the Prevena dressing system.

Negative pressure wound therapy has been applied for many years to enhance healing of a variety of open wounds including pressure wounds, diabetic ulcers, venous stasis ulcers, open infected surgical to traumatic wounds and burns with variable success. The treatment is based on evenly distributed local negative pressure applied to the wound surface. The open wound is filled with a sponge and covered with an occlusive dressing which is then connected by means of a set of suction tubes to a device which applies negative pressure on the surface of the wound that can be adjusted either cyclically or continuously. The fluid from the wound is collected into a container. The benefits of negative pressure wound therapy have been reported to include removal of infectious material, reduction in edema and improved perfusion to tissue.

The success of negative pressure wound therapy with open wounds has been extrapolated to intact surgical incisions. Recently a negative pressure wound therapy dressing has been developed for use over closed surgical incisions.

The investigators aim to study the ability of a negative pressure wound therapy dressing to prevent wound complications after vascular surgery involving incisions in the groin.

The aim of this study is to compare the Prevena dressing system to standard surgical dressing in patients undergoing leg bypass surgery or femoral endarterectomy with or without patch angioplasty involving the common femoral artery and/or profunda and/or proximal superficial femoral artery. The index groin may have undergone prior procedures (may be inflow or outflow for existing grafts), but the patient must have fully healed from the prior operation. May include patients with concomitant proximal and/or distal peripheral vascular intervention. The patch may be autogenous venous or arterial or prosthetic material such as bovine pericardium, dacron or polytetrafluoroethylene (PTFE) as well as bilateral femoral endartectomies are eligible for enrollment. The right and left groin incision would be randomized to the same dressing which is consistent with routine clinical practice. for vascular disease involving their legs in a multicenter randomized trial. All other aspects of the procedure are the part of standard vascular surgery practice. Patients undergoing vascular surgery with an incision in the groin will be treated with a standard gauze dressing or the Prevena wound management system which will be applied in the operating room and left on the wound for 5-7 days. Follow-up visits to assess the surgical wound are already standard of care. The two groups will be compared based on the primary and secondary endpoints listed in these documents. Quality of life will be compared by a patient survey and a cost analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Patient undergoing vascular surgery that would include a groin incision as a standard part of the operation. Infrainguinal bypass including femoral popliteal/tibial/pedal artery bypass with autogenous or prosthetic conduit.
3. femoral endarterectomy with or without patch angioplasty involving the common femoral artery and/or profunda and/or proximal superficial artery. The index groin may have undergone prior procedures (may be inflow or outflow for existing grafts), but the patient must have fully healed from the prior operation. May include patients with concomitant proximal and/or distal peripheral vascular intervention. The patch may be autogenous venous or arterial or prosthetic material such as bovine pericardium, dacron or polytetrafluoroethylene (PTFE). Bilateral femoral endarterectomies are eligible for enrollment. The right and left groin incision would be randomized to the same dressing which is consistent with routine clinical practice.
4. Willing to comply with protocol, attend follow-up appointments, complete all study assessments, and provide written informed consent.

Exclusion Criteria:

1. Any groin incision on index leg within 12 weeks prior to treatment initiation.
2. Infrainguinal bypass without a groin incision including popliteal-tibial or pedal bypass.
3. Supra inguinal procedures such as open or endovascular abdominal aortic aneurysm repair or aorto-femoral/bi-femoral bypass for occlusive disease.
4. Undergoing current chemotherapy or radiation therapy.
5. Pregnancy or lactation.
6. Inability or refusal to provide informed consent.
7. Patients who received an investigational drug for peripheral arterial disease within 4 weeks of screening or who participated in another non-observational clinical trial in the prior 30 days.
8. Surgical incision in the groin without primary closure including previously open or infected wounds.
9. Sensitivity or allergy to silver.
10. Prior enrollment in this randomized controlled trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be a composite endpoint of surgical site infection as per Center for Disease Control definition, major wound non-infectious complications, or graft infection within 30 days of surgery. | 30 days

SECONDARY OUTCOMES:
surgical site infection alone at 30 days | 30 days
patient satisfaction as assessed by quality of life survey | 30 days
total costs including outpatient costs to 30 days postoperatively | 30 days
length of index hospital stay and any readmission for wound complications | 30 days
major adverse limb event (MALE) or postoperative death (POD). MALE includes above-ankle amputation of the index limb or major reintervention | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Bertges, MD, Principal Investigator — University of Vermont Medical Center
Locations (5):
- United States (5):
  - Maine Medical Center, Portland, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Vermont Medical Center, Burlington, Vermont

REFERENCES:
- [Background] Stewart AH, Eyers PS, Earnshaw JJ. Prevention of infection in peripheral arterial reconstruction: a systematic review and meta-analysis. J Vasc Surg. 2007 Jul;46(1):148-55. doi: 10.1016/j.jvs.2007.02.065. PMID 17606135
- [Background] Bandyk DF. Vascular surgical site infection: risk factors and preventive measures. Semin Vasc Surg. 2008 Sep;21(3):119-23. doi: 10.1053/j.semvascsurg.2008.05.008. PMID 18774446
- [Background] Kalish JA, Farber A, Homa K, Trinidad M, Beck A, Davies MG, Kraiss LW, Cronenwett JL; Society for Vascular Surgery Patient Safety Organization Arterial Quality Committee. Factors associated with surgical site infection after lower extremity bypass in the Society for Vascular Surgery (SVS) Vascular Quality Initiative (VQI). J Vasc Surg. 2014 Nov;60(5):1238-1246. doi: 10.1016/j.jvs.2014.05.012. Epub 2014 Jun 20. PMID 24953898
- [Background] Khuri SF, Daley J, Henderson W, Hur K, Demakis J, Aust JB, Chong V, Fabri PJ, Gibbs JO, Grover F, Hammermeister K, Irvin G 3rd, McDonald G, Passaro E Jr, Phillips L, Scamman F, Spencer J, Stremple JF. The Department of Veterans Affairs' NSQIP: the first national, validated, outcome-based, risk-adjusted, and peer-controlled program for the measurement and enhancement of the quality of surgical care. National VA Surgical Quality Improvement Program. Ann Surg. 1998 Oct;228(4):491-507. doi: 10.1097/00000658-199810000-00006. PMID 9790339
- [Background] Ozaki CK, Hamdan AD, Barshes NR, Wyers M, Hevelone ND, Belkin M, Nguyen LL. Prospective, randomized, multi-institutional clinical trial of a silver alginate dressing to reduce lower extremity vascular surgery wound complications. J Vasc Surg. 2015 Feb;61(2):419-427.e1. doi: 10.1016/j.jvs.2014.07.034. Epub 2014 Aug 28. PMID 25175629
- [Background] Nguyen LL, Brahmanandam S, Bandyk DF, Belkin M, Clowes AW, Moneta GL, Conte MS. Female gender and oral anticoagulants are associated with wound complications in lower extremity vein bypass: an analysis of 1404 operations for critical limb ischemia. J Vasc Surg. 2007 Dec;46(6):1191-1197. doi: 10.1016/j.jvs.2007.07.053. PMID 18154995
- [Background] Matatov T, Reddy KN, Doucet LD, Zhao CX, Zhang WW. Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. Epub 2013 Jan 9. PMID 23312938
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- See also: Prevention of infection in peripheral arterial reconstruction: a systematic review and meta-analysis. J Vasc Surg. 2007 Jul;46(1):148-55. Review. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Stewart+AH%2C+Eyers+PS%2C+Earnshaw+JJ.+Prevention+of+infection+in+peripheral+arterial+reconstruction%3A+a+systematic+review+and+meta-analysis.+J+Vasc+Surg.+2007+Jul%3B46(1)%3A148-55.+Review.
- See also: Vascular surgical site infection: risk factors and preventive measures. Semin Vasc Surg. 2008 Sep;21(3):119-23. doi: 10.1053/j.semvascsurg.2008.05.008. Review. — http://www.ncbi.nlm.nih.gov/pubmed/18774446
- See also: Factors associated with surgical site infection after lower extremity bypass in the — http://www.ncbi.nlm.nih.gov/pubmed/24953898
- See also: The Department of Veterans Affairs' NSQIP: the first national, validated, outcome-based, risk-adjusted, and peer-controlled program for the measurement and enhancement of the quality of surgical care. National VA Surgical Quality Improvement Program. Ann — http://www.ncbi.nlm.nih.gov/pubmed/9790339
- See also: Prospective, randomized, multi-institutional clinical trial of a silver alginate dressing to reduce lower extremity vascular surgery wound complications. J Vasc Surg. 2015 Feb;61( — http://www.ncbi.nlm.nih.gov/pubmed/25175629
- See also: Female gender and oral anticoagulants are associated with wound complications in lower extremity vein bypass: an analysis of 1404 operations for critical limb ischemia. J Vasc — http://www.ncbi.nlm.nih.gov/pubmed/18154995
- See also: Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. E — http://www.ncbi.nlm.nih.gov/pubmed?term=%22Journal+of+vascular+surgery%22%5BJour%5D+AND+matatov%5Bauthor%5D&cmd=detailssearch